CLINICAL TRIAL: NCT04918238
Title: Effect of Muscle Energy Techniques on Functional Abilities in Patients With Discogenic Unilateral Sciatica
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Horus University (Other)
Responsible Party: Principal Investigator, Basem Muhammad Khalefa, Principal Investigator, Horus University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Basem_MSc
Record Dates: First submitted 2021-06-02; First posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Sciatica; Low Back Pain
MeSH Terms: conditions — Sciatica; Low Back Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional treatment Arm (Active Comparator): All the participants will receive the conventional physical therapy protocol per session as following: Infrared radiation on the low back area for 15 minutes, Ultrasound waves (Digi sonic device) for 10 minutes on the trigger areas of the low back, Myofascial release of the thoracolumbar fascia, Stretching of the Paraspinal muscles and the hamstrings, Mobilization of the lumbar and thoracic spine from a prone lying position and strengthening of abdominal muscles, multifidus and transversal's abdominal muscle.
  Interventions: Other: Conventional program
- muscle energy technique arm (Experimental): Group A received muscle energy technique with lateral recumbent positioning along with Conventional Physiotherapy Program
  Interventions: Other: Conventional program; Other: Muscle energy technique

INTERVENTIONS:
Other: Conventional program — All the participants will receive the conventional physical therapy protocol per session as following: Infrared radiation on the low back area for 15 minutes, Ultrasound waves (Digi sonic device) for 10 minutes on the trigger areas of the low back, Myofascial release of the thoracolumbar fascia, Stretching of the Paraspinal muscles and the hamstrings, Mobilization of the lumbar and thoracic spine from a prone lying position and strengthening of abdominal muscles, multifidus and transversal's abdominal muscle.
Other: Muscle energy technique — The patient was in the lateral recumbent position on the side opposite to his, her side-bending dysfunction while the physiotherapist stood facing the subject. The physiotherapist monitored the lumbar area with one hand while with the other hand flexed the subject's knees and hips until the barrier was engaged at the vertebral segment being treated.
  Arms: muscle energy technique arm

SUMMARY:
The purpose of the study to investigate the effect of muscle energy techniques on functional abilities of patients with chronic discogenic unilateral sciatica and to explain it from a physiological and functional point of view

DETAILED DESCRIPTION:
Disability and emotional distress among patients with lumbar spondylosis has a negative impact on well-being. Anxiety and depression are common emotional problems among patients with LBP.

The experience of pain interferes with different aspects of the patient's life, negatively affecting their daily activities, physical and mental health, family and social relationships, and their interactions in the workplace.

This problem also affects the health care system and what is known as economic well-being, the strong burden associated with Chronic Pain not only deriving from healthcare costs but also from the loss of productivity and from compensatory payments to patients as a result of the disability that pain produces.

Movement research has vast implications for muscle energy techniques for individuals with chronic low back pain and sciatica, the thoracolumbar normal range of motion plays an essential role in transferring the body weight and performing daily activities. Poor spinal range of motion and tightness of paraspinal muscles have previously been noted in individuals with chronic low back pain and sciatica.

Most of the previous studies focused on dealing with chronic low back pain and sciatica through using different medications and physical therapy modalities for the symptoms such as TENS. Since muscle energy techniques can decrease the tension of the muscles of the lumbar spine and gives a real chance to improve the flexibility of those muscles which might inhibit the severity of sciatica with low costs so it's recommended to study its effect on the functional abilities of the patients so that it can be the main part of physical therapy rehabilitation protocol.

ELIGIBILITY:
Inclusion Criteria:

* History of sciatica for more than 12 weeks or has at least 3 episodes of intermittent sciatica, each last for morethan 1 week eitheraccompanied with low back pain during the 3 months before thestudy. Medically and radiologically diagnosed as discogenic chronic sciatica with mild to moderate disability according to modified Rolland and Morris scale.

  * Both males and females, aged from 25 to 40 years old.
  * Be able to understand and follow the instructions during testing and treatment procedures

Exclusion Criteria:

* Fracture of pelvis, spine or lower extremities.

  * Hospitalization for severe trauma.
  * Peripheral neuropathy of diabetes or any other autoimmune disease.
  * Systematic autoimmune disease such as rheumatoid arthritis, systematic lupus
  * People with red flags such as cancer or severe osteoporosis.
  * Symptoms provoked while doing active hip joint extension and abduction.
  * Previous surgery to the lumbar spine, abdomen, pelvis, or hip.
  * Any contraindication for exercise therapy (e.g. uncontrolled hypertension, previous myocardial infarction, cardiovascular disease, peripheral vascular disease, respiratory disorders).
  * Any pain originated because of SI pathology.
  * Menstruation during testing days.
  * Individuals incapable of understanding and answering the Questionnaire.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) | "through study completion, an average of 2 months"
  Change from baseline Pain and at 2 months
Oswestry disability index scale | "through study completion, an average of 2 months"
  Change from baseline disability and at 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient clinic - Faculty of Physical Therapy - Horus University, Damietta, Egypt

IPD SHARING:
Plan to Share IPD: No